CLINICAL TRIAL: NCT00099112
Title: Transcriptional Profiling of the Epidermal Response to Solar-Simulated Ultraviolet Radiation
Brief Title: Effect of Solar-Simulated Ultraviolet Radiation on Gene Expression in Unprotected and Sunscreen-Protected Skin of Healthy Adults With Fitzpatrick Skin Type II
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000357437; NCI-04-C-0120; NCT00077740 (obsolete NCT alias)
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2005-11

CONDITIONS: Non-melanomatous Skin Cancer; Precancerous Condition
Keywords: basal cell carcinoma of the skin; squamous cell carcinoma of the skin; actinic keratosis
MeSH Terms: conditions — Precancerous Conditions; Carcinoma, Basal Cell; Keratosis, Actinic | interventions — Microarray Analysis; Biopsy

INTERVENTIONS:
Genetic: microarray analysis
Procedure: biopsy
Procedure: evaluation of cancer risk factors

SUMMARY:
RATIONALE: Testing of skin that has been exposed to artificial sunlight may help in understanding the genetic processes involved in the development of skin cancer.

PURPOSE: This trial is studying the effect of solar-simulated ultraviolet radiation on skin with or without sunscreen in healthy adults with skin that burns easily after only slight tanning during sun exposure.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the global gene expression profiles in epidermal tissue of healthy fair-skinned adults with Fitzpatrick skin type II after exposure to known doses of solar-simulated ultraviolet radiation (ssUVR) (UVA).
* Determine the ability of an FDA-standardized sunscreen to alter ssUVR-induced transcription profiles in vivo in these participants.
* Determine whether the transcriptional profiles of keratinocytes exposed to UVR in cell culture are comparable to the profiles of keratinocytes in skin after similar levels of UVR exposure.

OUTLINE: This is a pilot, dose-response study followed by an in vivo transcriptional profiling study in 2 different groups.

* Pilot study (verification of ultraviolet radiation dose response): Participants are initially exposed to solar-simulated ultraviolet radiation (ssUVR) (UVA) on the back to determine the minimum erythema dose (MED). Between 22-24 hours after exposure, participants undergo shave biopsy from each of the 9 UV exposure sites and 1 unexposed skin site.
* Group 1 (determination of ssUVR and UVA in vivo transcriptional profiles): On day 1, participants are initially exposed to ssUVR on the back to determine the MED. On day 2, participants are exposed to ssUVR (3 sites) and UVA (3 sites) at the MED on the buttocks. Between 22-24 hours after exposure (day 3), participants undergo shave biopsy from each of the 6 UV exposure sites and 2 unexposed skin sites.
* Group 2 (determination of sunscreen-protected in vivo transcriptional profiles): On day 1, participants are initially exposed to ssUVR on the back to determine the MED. On day 2, participants are exposed to ssUVR on unprotected skin (3 sites) and sunscreen-protected skin (3 sites) at the MED on the buttocks. Between 22-24 hours after exposure (day 3), participants undergo shave biopsy from each of the 6 UV exposure sites and 2 unexposed skin sites.

Biopsies from all participants are analyzed by microarray analysis. One of the unexposed epidermal samples is used for primary keratinocyte culture.

PROJECTED ACCRUAL: A total of 6-56 participants (6 for the pilot study and 50 [25 per group] for transcriptional profiling) will be accrued for this study within 2 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy, fair-skinned adults
* Fitzpatrick skin type II by history and physical exam

  * Skin easily burns, and tans only slightly, after sun exposure
* Test site for solar-simulated ultraviolet radiation exposure (buttocks) devoid of sunburn, suntan, scars, active dermal lesions, and uneven skin tones

  * Nevi allowed at physician discretion
  * Excess hair must be clipped or shaved
* No prior nonmelanoma skin cancer, melanoma, or dysplastic nevi

PATIENT CHARACTERISTICS:

Age

* 18 to 45

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No prior malignancy
* No prior phototoxic, photoallergic, or other abnormal responses to sunlight
* No prior allergic reaction to sunscreen or lidocaine
* No underlying disease that is known to cause immunosuppression (e.g., HIV, cancer, or post-organ transplantation)
* No situation that would preclude study compliance
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 6 months since prior topical or systemic medication producing abnormal sunlight responses
* No concurrent medications with > 1% incidence of sun-related toxic effects
* No concurrent medications associated with abnormal light response
* No concurrent immunosuppressants
* No other concurrent ultraviolet radiation (e.g., sunlight or tanning bed) to the epidermal test site

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2004-02

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C. Vogel, MD, Study Chair — NCI - Dermatology Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States